CLINICAL TRIAL: NCT02872389
Title: Power Spectral Analysis of the Electroencephalogram During Equi-MAC Sevoflurane vs. Desflurane Anesthesia: A Randomized Controlled Trial
Brief Title: Power Spectral Analysis of EEG During Equi-MAC Inhalation Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Kyoung-Ho Ryu, MD, Clinical assistant professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KBSMC 2016-07-033
Record Dates: First submitted 2016-08-10; First posted 2016-08-19 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Anesthesia
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Experimental): Anesthesia was maintained with sevoflurane.
  Interventions: Drug: Sevoflurane
- Desflurane (Experimental): Anesthesia was maintained with desflurane.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Anesthesia was maintained with sevoflurane in patients undergoing arthroscopic knee surgery under general anesthesia. End-tidal concentration of sevoflurane was maintained at age-corrected 1 minimum alveolar concentration throughout the study period.
  Other Names: SEVO
  Arms: Sevoflurane
Drug: Desflurane — Anesthesia was maintained with desflurane in patients undergoing arthroscopic knee surgery under general anesthesia. End-tidal concentration of desflurane was maintained at age-corrected 1 minimum alveolar concentration throughout the study period.
  Other Names: DES
  Arms: Desflurane

SUMMARY:
The purpose of this clinical trial is to compare hypnotic effect of sevoflurane and desflurane at equal minimum alveolar concentrations using power spectral analysis of the electroencephalogram.

DETAILED DESCRIPTION:
Volatile anesthetics vary in their relative hypnotic potency. Recent studies demonstrated that equi-minimum alveolar concentration of various volatile anesthetic agents may produce different spectral entropy or bispectral index values. However, there were no studies that demonstrate the difference of hypnotic potency using power spectral analysis of electroencephalographic signals (e.g., spectral edge frequency 95%, total power, % value of each bandage). The purpose of this clinical trial is to compare hypnotic effect of sevoflurane and desflurane at equal minimum alveolar concentrations using power spectral analysis of the electroencephalogram.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing arthroscopic knee surgery under general anesthesia using volatile anesthetics
* patients with american society of anesthesiologist physical status I, II
* patients aged 19-65 years
* patients obtaining written informed consent

Exclusion Criteria:

* patients with a history of any psychiatric or neurological disease
* patients who had received any medication affecting the central nervous system
* patients who had received medication affecting the sympathetic or parasympathetic nervous systems
* patients undergoing tracheal intubation for airway management
* pregnant women

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-06 (Actual)

PRIMARY OUTCOMES:
Spectral edge frequency 95% value | During about 30 min study period
  EEG variables were measured after meeting steady-state anesthesia of 1 MAC.

SECONDARY OUTCOMES:
Bispectral index | During about 30 min study period
  Bispectral index measurements were made after meeting steady-state anesthesia of 1 MAC.

CONTACTS AND LOCATIONS:
Overall Officials: Kyoungho Ryu, M.D., Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided